CLINICAL TRIAL: NCT02922855
Title: Incentives for Primary Care Use: A Randomized Controlled Trial in a Safety Net Setting
Brief Title: Incentives for Primary Care Use in a Safety Net Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HM20000002; 1R01HS022534 (AHRQ)
Record Dates: First submitted 2016-09-28; First posted 2016-10-04 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Health Care Utilization; Primary Care Physician; Uninsured
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Contemporaneous Control (No Intervention): This group is our 'usual care' control group. They were not contacted for an interview and were not offered an incentive to visit their primary care physician.
- $0 group (Active Comparator): This group completed a baseline interview but was not offered any incentive if they visited their primary care physician.
  Interventions: Behavioral: 0 dollars group
- $25 group (Experimental): This group completed a baseline interview and was offered $25 they visited their primary care physician within 6 months.
  Interventions: Behavioral: 25 dollars group
- $50 group (Experimental): This group completed a baseline interview and was offered $50 they visited their primary care physician within 6 months.
  Interventions: Behavioral: 50 dollars group

INTERVENTIONS:
Behavioral: 0 dollars group — Those assigned to the $0 group will not receive an incentive for visiting their PCP.
  Arms: $0 group
Behavioral: 50 dollars group — Those assigned to the $50 group will receive $50 if they visit their PCP within 6 months of study enrollment.
  Arms: $50 group
Behavioral: 25 dollars group — Those assigned to the $25 group will receive $25 if they visit their PCP within 6 months of study enrollment.
  Arms: $25 group

SUMMARY:
A randomized controlled trial (RCT) of incentives for an initial primary care visit within 6 months of enrollment in a health care coverage program. Study subjects are drawn from a low-income adult population that gains coverage and access to community-based primary care services under a program administered by an academic safety-net hospital. The investigators will offer financial incentives to encourage an initial primary care visit within 6 months of enrollment and evaluate whether the primary care visit altered subsequent health seeking behavior and influenced patient satisfaction and other outcomes such as self-reported health status.

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) of incentives for an initial primary care visit within 6 months of enrollment in a health care coverage program. Study subjects are drawn from a low-income adult population that gains coverage and access to community-based primary care services under a program administered by an academic safety-net hospital. The investigators will offer financial incentives to encourage an initial primary care visit within 6 months of enrollment and evaluate whether the primary care visit altered subsequent health seeking behavior and influenced patient satisfaction and other outcomes such as self-reported health status.

Incentives should steer patients in their decision to seek primary care, reduce barriers to care, and ultimately improve patient health and reduce utilization and costs through their relationship with a PCP. This study is the first of its kind to incentivize low-income patients. This population has the greatest need for health care and exerts the greatest pressure on the United States' safety net system. Furthermore, the safety net population is the target of policies such as Medicaid eligibility expansions, yet urban safety net patients are largely understudied. These patients are rarely given the opportunity to participate in research, and when they are the subjects of measures to reduce health care utilization, they are the subject of policies using negative incentives such as those that introduce cost sharing for using ED services.1 Alternatively, safety net providers invest in case management systems to reduce utilization. The proposed study is a departure from prior measures to reduce utilization among low-income patients by focusing on patients and using positive incentives. The study borrows from the principles of behavioral economics to motivate patients towards primary care utilization. Once in the primary care system, The investigators will test whether primary care contact reduces more expensive forms (e.g., inpatient, ED) of health care.

The investigators will compare outcomes of patients assigned in the highest incentive group ($50) to patients assigned to the modest incentive group ($25) and to patients assigned to usual care (no incentive, but assignment to a PCP). The investigators will also compare incentive patients ($50, $25) to a contemporaneous group of patients that enroll in the safety net clinic at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Adults between ages 21-64 years
* No prior enrollment in VCC for the past 12 months
* English or Spanish speaking, and
* Can be contacted by mail and telephone (preferably) or willing to be interviewed in person.

Exclusion Criteria:

* Unable to be contacted by phone/mail
* Cannot provide consent
* No longer located in catchment area

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1228 (Actual)
Dates: Start 2014-01; Primary Completion 2016-11-08 (Actual); Study Completion 2016-11-08 (Actual)

PRIMARY OUTCOMES:
The number of Primary Care Physician visits will be assessed using medical claims record data. | This will be assessed in the 6 months following study enrollment.
  The number of primary care visits to a primary care physician will be collected from medical claims record data.

SECONDARY OUTCOMES:
The time to a Primary Care Physician will be assessed using medical claims record data. | This will be assessed in the 6 months following study enrollment.
  The time to a primary care visits to a primary care physician will be collected from dates available in the medical claims record data.

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Bradley, Phd, Principal Investigator — PI

IPD SHARING:
Plan to Share IPD: No